CLINICAL TRIAL: NCT05450679
Title: The Predictive Value of Cervical Paraspinal Muscle Twitching During Motor Stimulation Testing on Cervical Facet Joint Radiofrequency Ablation Outcomes
Brief Title: Cervical Paraspinal Muscle Twitching and Cervical Facet Radiofrequency Ablation Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00323880
Record Dates: First submitted 2022-07-05; First posted 2022-07-11 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Cervical Facet Joint Pain; Chronic Pain; Neck Pain
Keywords: facet arthropathy; cervicalgia; radiofrequency ablation
MeSH Terms: conditions — Chronic Pain; Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervical Radiofrequency Ablation (RFA)-treated group: Only patients who have already been deemed candidates by their primary pain physician for cervical RFA will be recruited to the study. During the cervical RFA procedure, all patients will undergo sensory and motor stimulation testing prior to receiving radiofrequency lesioning, which is a standard and recommended practice.
  Interventions: Procedure: Cervical Radiofrequency Ablation (RFA)

INTERVENTIONS:
Procedure: Cervical Radiofrequency Ablation (RFA) — During the cervical RFA procedure, all patients will undergo sensory and motor stimulation testing prior to receiving radiofrequency lesioning, which is a standard and recommended practice.
  During the motor stimulation testing step, the pain physicians performing the procedure will assess the presence or absence of cervical paraspinal muscle twitching by using a standardized grading scale (per radiofrequency electrode: 0 = no twitches observed or palpated; 1 = twitches palpated but not observed; 2 = twitches observed and palpated at 1-2 levels; 3 = twitches observed at > 2 levels). A total score and a weighted score (total score divided by the number of radiofrequency lesion sites), will be recorded for each patient, and the RFA procedure will be completed per usual practice.
  RFAs will be performed in the usual manner and as per "standard of care." Providers will not use any new or experimental devices to perform the RFA.

SUMMARY:
The investigators aim to determine whether cervical paravertebral muscle twitching during motor testing as part of performing cervical RFAs is associated with a greater likelihood of treatment success, and greater magnitude or duration of analgesia. The investigators propose a straightforward grading scale based on visual and tactile information readily available during RFA procedures as part of routine practice (per radiofrequency electrode: 0 = no twitches palpated or observed; 1 = twitches palpated but not observed; 2 = twitches palpated and observed at 1-2 levels; 3= twitches palpated and observed at >2 levels). If a higher weighted score (total score divided by number of radiofrequency lesion sites) correlates with a greater likelihood of treatment success, or magnitude or duration of analgesia following cervical RFA, cervical paraspinal muscle twitching may serve as a readily obtainable prognostic factor (marker) for effectiveness.

DETAILED DESCRIPTION:
Approximately 60 patients with cervical facet arthropathy who are undergoing cervical radiofrequency ablation (RFA) will be recruited for this study. Only patients who have already been deemed candidates by their primary pain physician for cervical RFA (e.g. > 50% relief from a diagnostic cervical medial branch block) will be recruited. During the cervical RFA procedure, all patients will undergo sensory and motor stimulation testing prior to receiving radiofrequency lesioning, which is a standard and recommended practice. The investigators will align the electrodes to optimize sensory testing.

During the motor stimulation testing step, the pain physicians performing the procedure (e.g. attending, fellows, residents, etc.) will assess the presence or absence of cervical paraspinal muscle twitching by using a standardized grading scale (per radiofrequency electrode: 0 = no twitches observed or palpated; 1 = twitches palpated but not observed; 2 = twitches observed and palpated at 1-2 levels; 3 = twitches observed at > 2 levels). A total score and a weighted score (total score divided by the number of radiofrequency lesion sites), will be recorded for each patient, and the RFA procedure will be completed per usual practice.

The interventional procedure used in this study (radiofrequency ablation) will be performed in the usual manner and as per "standard of care." The use of the grading scale described above to assess the presence/absence and magnitude of cervical paraspinal muscle twitching will be unique to this research study.

The investigators will also obtain the following data immediately pre-procedurally, from electronic health record review and also a standardized set of questionnaires provided to study participants:

* Information routinely obtained as standard practice: age, sex, average and worst neck pain score over the past week on numeric rating scale (NRS), percent pain relief from diagnostic block, duration of pain, inciting event, MRI findings if available, obesity (defined as BMI > 30), smoking, co-existing pain conditions, co-existing psychiatric conditions, and potential sources of secondary gain (e.g. worker's compensation claim, ongoing litigation, etc.)
* Information obtained as part of the research study: Neck Disability Index (NDI) score, Athens Insomnia Scale (AIS) score, Hospital Anxiety and Depression Scale (HADS) scores.

At a 1-month post-procedural follow-up timepoint, the investigators will obtain the following data, from electronic health record review and also a standardized set of questionnaires provided to study participants:

* Information routinely obtained as standard practice: categorical binary outcome (positive outcome defined as >/= 2-point decrease in average neck pain score coupled with PGIC score >/= 5/7) analgesic medications and doses; status of medication reduction (yes or no); average and worst NRS pain score over the past week; description of any procedural complications
* Information obtained as part of the research study: NDI, AIS, and HADS scores; Patient Global Impression of Change Scale (PGIC) score
* Exiting the trial: patients may choose to exit the study at any time for any reason. A patient will exit the study to receive alternative care if the patient reports a PGIC score <5 or < 2-point reduction in average NRS pain score. This would indicate that the RFA treatment was unsuccessful.

At a 3-month post-procedural follow-up timepoint, the investigators will obtain the following data, from electronic health record review and also a standardized set of questionnaires provided to study participants:

* Information routinely obtained as standard practice: categorical binary outcome, analgesic medications and doses; status of medication reduction (yes or no); average and worst NRS pain score over the past week; description of any procedural complications
* Information obtained as part of the research study: NDI, AIS, and HADS scores; Patient Global Impression of Change Scale (PGIC) score on 7-point Likert scale
* Exiting the trial: patients may choose to exit the study at any time for any reason. A patient will exit the study to receive alternative treatment if the patient reports a PGIC score <5 or < 2-point reduction in average NRS pain score. This would indicate that the analgesic and functional benefit of the RFA procedure has now been exhausted.

At a 6-month post-procedural follow-up timepoint, the investigators will obtain the following data, from electronic health record review and also a standardized set of questionnaires provided to study participants:

* Information routinely obtained as standard practice: binary categorical outcome, analgesic medications and doses; status of medication reduction (yes or no); average and worst NRS pain score over the past week; description of any procedural complications
* Information obtained as part of the research study: NDI, AIS, and HADS scores; Patient Global Impression of Change Scale (PGIC) score
* Exiting the trial: All patients who remain in the study will exit at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Cervical facet arthropathy based on history and physical exam (e.g. axial cervical neck pain, paraspinal tenderness, no pain referral below the ipsilateral shoulder)
* Radiologic evidence of cervical pathology consistent with symptoms if MRI is available
* Pain duration of greater than 3 months
* Obtained 50% or greater pain relief from at least 1 diagnostic cervical medial branch block of the identical medial branch nerves targeted for RFA

Exclusion Criteria:

* Untreated coagulopathy
* Signs or symptoms of cervical myelopathy
* Signs or symptoms of cervical radiculitis/radiculopathy
* Allergic reactions to local anesthetics
* Serious psychiatric disorder (e.g. uncontrolled or refractory depression) that might preclude optimal outcome
* Poorly controlled medical condition (e.g. pacemaker that cannot be switched off, unstable angina)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only patients who have already been deemed candidates by their primary pain physician for a cervical radiofrequency ablation (RFA) (e.g. >/= 50% relief from a diagnostic cervical medial branch block) will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Categorical number of participants with treatment success or failure | 3 months
  Definition of success: a >/= 2-point decrease in average neck pain (measured over the past week) coupled with a score of >/= 5/7 on a patient global impression of change (PGIC) scale where 1= "no change or worsened symptoms", 5= "moderately better, a slight but noticeable change", and 7= "a great deal better."

SECONDARY OUTCOMES:
Categorical number of participants with treatment success or failure | 1 month
  Definition of success: a >/= 2-point decrease in average neck pain (measured over the past week) coupled with a score of >/= 5/7 on a patient global impression of change (PGIC) scale where 1= "no change or worsened symptoms", 5= "moderately better, a slight but noticeable change", and 7= "a great deal better."
Categorical number of participants with treatment success or failure | 6 months
  Definition of success: a >/= 2-point decrease in average neck pain (measured over the past week) coupled with a score of >/= 5/7 on a patient global impression of change (PGIC) scale where 1= "no change or worsened symptoms", 5= "moderately better, a slight but noticeable change", and 7= "a great deal better."
Average neck pain score | 1 month
  Pain scores measured on 0-10 numeric rating scale (NRS)
Average neck pain score | 3 months
  Pain scores measured on 0-10 numeric rating scale (NRS)
Average neck pain score | 6 months
  Pain scores measured on 0-10 numeric rating scale (NRS)
Worst neck pain score | 1 month
  Pain scores measured on 0-10 numeric rating scale (NRS)
Worst neck pain score | 3 months
  Pain scores measured on 0-10 numeric rating scale (NRS)
Worst neck pain score | 6 months
  Pain scores measured on 0-10 numeric rating scale (NRS)
Functional outcome as measured using the Neck disability index (NDI) | 1 month
  Neck disability index (NDI) score (0-100%, higher numbers indicate poorer function)
Functional outcome as measured using the Neck disability index (NDI) | 3 months
  Neck disability index (NDI) score (0-100%, higher numbers indicate poorer function)
Functional outcome as measured using the Neck disability index (NDI) | 6 months
  Neck disability index (NDI) score (0-100%, higher numbers indicate poorer function)
Sleep quality as assessed by the Athens Insomnia Scale (AIS) | 1 month
  Athens Insomnia Scale (AIS) score (0-24, with higher scores indicate greater dysfunction)
Sleep quality as assessed by the Athens Insomnia Scale (AIS) | 3 months
  Athens Insomnia Scale (AIS) score (0-24, with higher scores indicate greater dysfunction)
Sleep quality as assessed by the Athens Insomnia Scale (AIS) | 6 months
  Athens Insomnia Scale (AIS) score (0-24, with higher scores indicate greater dysfunction)
Mood and anxiety as assessed by the Hospital anxiety and depression scale (HADS) | 1 month
  Hospital anxiety and depression scale (HADS) score (Depression and anxiety scored from 0-21 with higher scores indicating greater depression and anxiety)
Mood and anxiety as assessed by the Hospital anxiety and depression scale | 3 months
  Hospital anxiety and depression scale (HADS) score (Depression and anxiety scored from 0-21 with higher scores indicating greater depression and anxiety)
Mood and anxiety as assessed by the Hospital anxiety and depression scale | 6 months
  Hospital anxiety and depression scale (HADS) score (Depression and anxiety scored from 0-21 with higher scores indicating greater depression and anxiety)
Medication reduction as assessed by follow-up visit or telephone call, and Prescription Drug Monitoring Program data review | 1 month
  Defined as cessation of a non-opioid analgesic or > 20% decrease in pre-existing opioid consumption
Medication reduction as assessed by follow-up visit or telephone call, and Prescription Drug Monitoring Program data review | 3 months
  Defined as cessation of a non-opioid analgesic or > 20% decrease in pre-existing opioid consumption
Medication reduction as assessed by follow-up visit or telephone call, and Prescription Drug Monitoring Program data review | 6 months
  Defined as cessation of a non-opioid analgesic or > 20% decrease in pre-existing opioid consumption
Procedural complications | Any time point up to the 6-month post-procedural follow-up visit or up to the patient exiting the trial (whichever occurs first)
  Any reported adverse events or complications directly related to the cervical radiofrequency ablation (RFA) procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wang, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.

REFERENCES:
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] Aprill C, Bogduk N. The prevalence of cervical zygapophyseal joint pain. A first approximation. Spine (Phila Pa 1976). 1992 Jul;17(7):744-7. doi: 10.1097/00007632-199207000-00003. PMID 1502636
- [Background] Manchikanti L, Singh V, Rivera J, Pampati V. Prevalence of cervical facet joint pain in chronic neck pain. Pain Physician. 2002 Jul;5(3):243-9. PMID 16902649
- [Background] Schaerer JP. Radiofrequency facet rhizotomy in the treatment of chronic neck and low back pain. Int Surg. 1978 Sep-Dec;63(6):53-9. PMID 155664
- [Background] Lord SM, Barnsley L, Wallis BJ, McDonald GJ, Bogduk N. Percutaneous radio-frequency neurotomy for chronic cervical zygapophyseal-joint pain. N Engl J Med. 1996 Dec 5;335(23):1721-6. doi: 10.1056/NEJM199612053352302. PMID 8929263
- [Background] Huygen F, Kallewaard JW, van Tulder M, Van Boxem K, Vissers K, van Kleef M, Van Zundert J. "Evidence-Based Interventional Pain Medicine According to Clinical Diagnoses": Update 2018. Pain Pract. 2019 Jul;19(6):664-675. doi: 10.1111/papr.12786. Epub 2019 May 2. PMID 30957944
- [Background] Hurley RW, Adams MCB, Barad M, Bhaskar A, Bhatia A, Chadwick A, Deer TR, Hah J, Hooten WM, Kissoon NR, Lee DW, Mccormick Z, Moon JY, Narouze S, Provenzano DA, Schneider BJ, van Eerd M, Van Zundert J, Wallace MS, Wilson SM, Zhao Z, Cohen SP. Consensus practice guidelines on interventions for cervical spine (facet) joint pain from a multispecialty international working group. Reg Anesth Pain Med. 2022 Jan;47(1):3-59. doi: 10.1136/rapm-2021-103031. Epub 2021 Nov 11. PMID 34764220
- [Background] Lord SM, McDonald GJ, Bogduk N. Percutaneous Radiofrequency Neurotomy of the Cervical Medial Branches. Neurosurgery Quarterly. 1998;8(4):288-308. doi:10.1097/00013414-199812000-00004
- [Background] MacVicar J, Borowczyk JM, MacVicar AM, Loughnan BM, Bogduk N. Cervical medial branch radiofrequency neurotomy in New Zealand. Pain Med. 2012 May;13(5):647-54. doi: 10.1111/j.1526-4637.2012.01351.x. Epub 2012 Mar 28. PMID 22458772
- [Background] Manchikanti L, Sanapati MR, Pampati V, Soin A, Atluri S, Kaye AD, Subramanian J, Hirsch JA. Update of Utilization Patterns of Facet Joint Interventions in Managing Spinal Pain from 2000 to 2018 in the US Fee-for-Service Medicare Population. Pain Physician. 2020 Mar;23(2):E133-E149. PMID 32214289
- [Background] International Spine Intervention Society. ISIS Practice Guidelines for Spinal Diagnostic and Treatment Procedures: 2nd Edition.; 2013. https://books.google.com/books/about/ISIS_Practice_Guidelines_for_Spinal_Diag.html?hl=&id=ikWhoAEACAAJ
- [Background] Cohen SP, Strassels SA, Kurihara C, Lesnick IK, Hanling SR, Griffith SR, Buckenmaier CC 3rd, Nguyen C. Does sensory stimulation threshold affect lumbar facet radiofrequency denervation outcomes? A prospective clinical correlational study. Anesth Analg. 2011 Nov;113(5):1233-41. doi: 10.1213/ANE.0b013e31822dd379. Epub 2011 Sep 14. PMID 21918166
- [Background] Dreyfuss P, Halbrook B, Pauza K, Joshi A, McLarty J, Bogduk N. Efficacy and validity of radiofrequency neurotomy for chronic lumbar zygapophysial joint pain. Spine (Phila Pa 1976). 2000 May 15;25(10):1270-7. doi: 10.1097/00007632-200005150-00012. PMID 10806505
- [Background] Koh JC, Kim DH, Lee YW, Choi JB, Ha DH, An JW. Relationship between paravertebral muscle twitching and long-term effects of radiofrequency medial branch neurotomy. Korean J Pain. 2017 Oct;30(4):296-303. doi: 10.3344/kjp.2017.30.4.296. Epub 2017 Sep 29. PMID 29123625